CLINICAL TRIAL: NCT04781959
Title: A Randomized, Multicenter Pragmatic Trial Comparing Bone Pain From a Single Dose of Pegfilgrastim to 5 Doses of Daily Filgrastim in Breast Cancer Patients Receiving Neoadjuvant/Adjuvant Chemotherapy (REaCT-5G)
Brief Title: A Randomized, Multicenter Pragmatic Trial Comparing Bone Pain From a Single Dose of Pegfilgrastim to 5 Doses of Daily Filgrastim in Breast Cancer Patients Receiving Neoadjuvant/Adjuvant Chemotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REaCT-5G
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Early-stage Breast Cancer
Keywords: Filgrastim; Pegfilgrastim
MeSH Terms: conditions — Breast Neoplasms | interventions — Filgrastim; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5 Days of Filgrastim (Active Comparator): Receive filgrastim subcutaneous injection once daily for five consecutive days starting 24-72 hours after chemotherapy.
  Interventions: Drug: Filgrastim
- Pegfilgrastim (Active Comparator): Receive pegfilgrastim as a single dose subcutaneous injection 24-72 hours after chemotherapy
  Interventions: Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Filgrastim — Receive filgrastim subcutaneous injection once daily for five consecutive days starting 24-72 hours after chemotherapy
  Other Names: Neupogen
  Arms: 5 Days of Filgrastim
Drug: Pegfilgrastim — Receive pegfilgrastim as a single dose subcutaneous injection 24-72 hours after chemotherapy
  Other Names: Neulasta
  Arms: Pegfilgrastim

SUMMARY:
REaCT-5G will compare bone pain from a single dose of Pegfilgrastim to 5 doses of daily filgrastim in breast cancer patients receiving neoadjuvant/adjuvant chemotherapy.

DETAILED DESCRIPTION:
The use of granulocyte colony-stimulating factors (G-CSF) significantly reduces febrile neutropenia (FN) risk and has helped maintain dose intensity and dose density when treating breast cancer with chemotherapy. This is crucial as survival outcomes are significantly impaired if dose intensity are reduced. National and international guidelines recommend the use of G-CSF as primary prophylaxis with most commonly used breast cancer chemotherapy regimens. Filgrastim (FIL) as a G-CSF that has been in use since the early 90s. Pegfilgrastim (PEG) is a long-acting, pegylated version of FIL that requires only one injection per chemotherapy cycle instead of daily FIL injections for 5 to 10 days per cycle. PEG and FIL both come at the potential cost of bone pain, the most common side effect. G-CSF related bone pain is often severe, leading to refusal or cancellation of G-CSF and early discontinuation of chemotherapy. We propose to perform a pragmatic, multicenter, open-label, randomized clinical trial to compare bone pain experienced by patients receiving either PEG or 5-day-FIL with neoadjuvant or adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with early-stage or locally-advanced breast cancer receiving neoadjuvant or adjuvant chemotherapy requiring primary febrile neutropenia prophylaxis with G-CSF
* Able to provide verbal consent
* Able to complete questionnaires in English or French

Exclusion Criteria:

* No access to pegfilgrastim or filgrastim prior to randomization
* Metastatic cancer
* Known hypersensitivity to filgrastim or pegfilgrastim or one of its components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Bone pain | 5 days after first G-CSF injection
  Bone pain over the first 5 days after the administration of G-CSF. The total measure of bone pain over the five days will be summarized by the area under the curve (AUC) based on a patient's daily pain score, starting after the first dose of G-CSF injection.

SECONDARY OUTCOMES:
Incidence of Febrile Neutropenia | 2.5 years after study initiation
  Number of times participants have Febrile neutropenia during chemotherapy treatment
Incidence of treatment-related hospitalizations | 2.5 years after study initiation
  Number of times participants have a treatment-related hospitalization
Incidence of chemotherapy alteration | 2.5 years after study initiation
  Number of times participants have a chemotherapy alteration including: dose delay, reduction and/or discontinuation
Incidence of chemotherapy-related mortality | 2.5 years after study initiation
  Number of times there is a chemotherapy-related mortality
Rate of G-CSF compliance as prescribed | 2.5 years after study initiation
  Number of times there is a G-CSF compliance
Differences in healthcare resource utilization | 2.5 years after study initiation
  Differences in healthcare resource utilization: number of emergency room visits, number of planned/unplanned provider clinic visits (including stretcher bay), patient-reported phone calls or email to patient support line or provider, and additional medication use or management strategies related to G-CSF side effects or efficacy
HR-QoL | 2.5 years after study initiation
  HR-QoL based on EQ-5D-5L
Cost-effectiveness | 2.5 years after study initiation
  Cost differences associated with prescribing Filgrastim and Pegfilgrastim
Patient G-CSF preference | 2.5 years after study initiation
  To survey patient preference in selection of G-CSF treatment before and after undergoing chemotherapy and G-CSF treatment
Study feasibility | 1 year after study initiation
  Interim analysis/feasibility. After the first year of study initiation, if study recruitment is less than 30% at one year (70 patients), or if there are unanticipated safety issues, a review of study conduct will be performed to consider stopping the study unless there are unexpected or exceptional reasons, or in the case of low recruitment, there is a plan to boost recruitment efforts

CONTACTS AND LOCATIONS:
Overall Officials: Terry Ng, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (2):
- Canada (2):
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario